CLINICAL TRIAL: NCT03812978
Title: Mobile Application for Improving Rehabilitation After Flexor Tendon Repair - A Randomized Controlled Multicenter Trial.
Brief Title: Mobile Application for Improving Rehabilitation After Flexor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marianne Arner, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FlexortendonsSOS2018
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Flexor Digitorum Profundus Injury
Keywords: "Flexor tendon rehabilitation"; "Smart-phone application"; "adherence"

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard treatment
- Intervention (Experimental): Standard treatment and intervention (Smart phone application)
  Interventions: Other: Smart phone application

INTERVENTIONS:
Other: Smart phone application — Smart phone application including exercise videos, push notifications for exercise, questions and answers, exercise diary.
  Arms: Intervention

SUMMARY:
Can a mobile application improve adherence, self-efficacy and range of motion after flexor tendon repair? A randomized controlled multicenter trial.

Aim Evaluate how the use of a mobile application will affect exercise adherence, range of motion and self-efficacy when compared to standard rehabilitation after flexor tendon repair. Method Multicenter randomized controlled trial. Patients with flexor tendon repair in zone I or II were included and rehabilitated with early active motion and followed 12 weeks post-surgery. Randomization was performed by a computer-generated concealed block to control (n=60) or intervention group (n=60). Both groups received standard rehabilitation according to early active motion. Intervention group also received a smart phone app including; exercise videos, push-notifications for exercise, exercise diary, written information on the surgery, rehabilitation, questions and answers. Evaluation was made at baseline, 2, 6- and 12-weeks after surgery. Primary outcome was physiotherapist rated adherence on the Sport Injury Adherence Scale (SIRAS). Secondary outcome was self-reported adherence, perceived self-efficacy, total Active range of motion (TAM) in the Proximal Interphalangeal (PIP) joint and Distal Interphalangeal (DIP) joint and perceived satisfaction with rehabilitation and information.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Own a mobile phone, fluent in Swedish,
* Suited for early active motion rehabilitation
* Injury to one or both of the flexor tendons in the a finger

Exclusion Criteria:

* concomitant fracture in the hand
* tendon injury to flexor pollicis longus.
* Extensor tendon injury in the same hand.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Sport injury adherence scale (SIRAS) | assessed at 2 weeks (totalt score range 3-15, higher value indicates better outcome)
  Physiotherapist rated adherence questionnaire
Sport injury adherence scale (SIRAS) | assessed at 6 weeks (totalt score range 3-15, higher value indicates better outcome)
  Physiotherapist rated adherence questionnaire

SECONDARY OUTCOMES:
Self reported adherence | assessed at 2 and 6 weeks (total score range 0-100,higher value indicates better outcome )
  Patient rated adherence questionnaire duration
Self reported adherence | assessed at 2 and 6 weeks (total score range 0-100,higher value indicates better outcome )
  Patient rated adherence questionnaire frequency
Self reported adherence | assessed at 2 and 6 weeks (total score range 0-100, higher value indicates better outcome)
  Patient rated adherence questionnaire quality
Athlet injury self efficacy questionnaire (AISEQ) | baseline, 2 and 6 weeks (Change over time)
  Patient reported self efficacy for rehabilitation
Range of motion | assessed at 12 weeks (range 0-240,higher value indicates better outcome )
  Total range of motion in the proximal interphalangeal and distal interphalangeal joints measured with a finger goniometer

OTHER OUTCOMES:
Perceived satisfaction with rehabilitation | at 12 weeks (range 0-100, higher value indicates better outcome)
  questions on a Likert scale regarding satisfaction of rehabilitation. "how do you perceive the rehabilitation after the operation?"
Perceived satisfaction with information | at 12 weeks (range 0-100, higher value indicates better outcome)
  questions on a Likert scale regarding satisfaction of information: "how do you perceive the information after the operation?"

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Arner, Phd, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Department of hand surgery, Skåne university hospital, Malmo
  - Department of hand surgery, University hospital Örebro, Örebro
  - Department of hand surgery, Södersjukshuset, Stockholm
  - Department of hand surgery, Uppsala university hospital, Uppsala